CLINICAL TRIAL: NCT00060541
Title: Evaluation and Treatment of Neurosurgical Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030164; 03-N-0164
Record Dates: First submitted 2003-05-07; First posted 2003-05-07 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-08-22

CONDITIONS: Neurologic Disorders
Keywords: Brain Tumor; Epilepsy; Pituitary Adenoma; Parkinson's Disease; Spinal Cord Tumor; Natural History
MeSH Terms: conditions — Nervous System Diseases; Brain Neoplasms; Epilepsy; Pituitary Neoplasms; Parkinson Disease; Spinal Cord Neoplasms | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients age 4 or older seeking care from, or being referred to the Surgical Neurology Branch for evaluation and management of neurosurgical conditions
  Interventions: Procedure: Laboratory tests; Procedure: Radiological exams

INTERVENTIONS:
Procedure: Laboratory tests
Procedure: Radiological exams

SUMMARY:
Objective: This protocol is designed to allow evaluation of participants neurosurgical disorders that receive care within the Surgical Neurology Branch. The participants will receive standard-of-clinical-care evaluation and treatment. The clinical data and samples generated during standard of care treatment will be collected as a part of this study.

Study Population: Participants 4 years of age and older with neurosurgical-related conditions seeking care from, or referred to the Surgical Neurology Branch for evaluation are eligible for this protocol.

Study Design: This is an observational study. Participants will receive standard-of- clinical-care evaluation and treatment for their neurosurgical condition. Clinical evaluation may include laboratory and radiological studies designed to aid in diagnosis or differential diagnosis of the participant s condition or to facilitate treatment. The evaluations may take place in the outpatient clinic areas or in the inpatient units. Some participants will receive standard-of-care medical or surgical treatment for their disorder. Clinical data, tissue samples or body fluids obtained during standard of care treatment, may be used for research. Additional genetic testing may be performed on subjects and their blood relatives if a genetic mechanism underlying the neurological disorder is suspected. Patients in this study may choose to consent to skin biopsies for research purposes, in which case they will sign an additional consent document for thesethis research procedure.

Outcome Measures: No additional research outcome measures will be tracked in this study, as this study is collecting data for potential future use. All outcomes will be those of standard clinical evaluation and treatment. A clinical and research database will be kept of patient s diagnosis, progression, and treatment. Clinical database information may be reported or be used in other studies.

DETAILED DESCRIPTION:
Objective: This protocol is designed to allow evaluation of participants neurosurgical disorders that receive care within the Surgical Neurology Branch. The participants will receive standard-of-clinical-care evaluation and treatment. The clinical data and samples generated during standard of care treatment will be collected as a part of this study.

Study Population: Participants 4 years of age and older with neurosurgical-related conditions seeking care from, or referred to the Surgical Neurology Branch for evaluation are eligible for this protocol.

Study Design: This is an observational study. Participants will receive standard-of- clinical-care evaluation and treatment for their neurosurgical condition. Clinical evaluation may include laboratory and radiological studies designed to aid in diagnosis or differential diagnosis of the participant s condition or to facilitate treatment. The evaluations may take place in the outpatient clinic areas or in the inpatient units. Some participants will receive standard-of-care medical or surgical treatment for their disorder. Clinical data, tissue samples or body fluids obtained during standard of care treatment, may be used for research. Additional genetic testing may be performed on subjects and their blood relatives if a genetic mechanism underlying the neurological disorder is suspected. Patients in this study may choose to consent to skin biopsies for research purposes, in which case they will sign an additional consent document for thesethis research procedure.

Outcome Measures: No additional research outcome measures will be tracked in this study, as this study is collecting data for potential future use. All outcomes will be those of standard clinical evaluation and treatment. A clinical and research database will be kept of patient s diagnosis, progression, and treatment. Clinical database information may be reported or be used in other studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participants must be age 4 and older.
  2. Participants must seek care from, or be referred to the Surgical Neurology Branch for evaluation and management of neurosurgical conditions (such as central nervous system tumors, peripheral nerve tumors, epilepsy, Parkinson s disease, movement disorders, Chiari syndrome, central nervous system malformations, and pain disorders)
  3. For adults: able to provide informed consent or having a legally-authorized representative to provide consent, if incapacitated
  4. For minors: a parent or legal guardian who is able to provide consent.

     For immediate blood relatives of subjects having genetic testing only:
  5. Blood relative of a subject who is suspected to have a genetic mechanism underlying their neurological disorder (for genetic testing only).

EXCLUSION CRITERIA:

1. Patients who are unable to undergo evaluation and treatment for a neurosurgical disorder

3.c. Participant Inclusion Criteria for the cohort with processing of biological samples only (for those subjects who are only having skin biopsies and/or saliva samples)

1. Participants must be age 4 and older.
2. Participants must seek care from or be referred to the Surgical Neurology Branch for evaluation and management of neurosurgical conditions (such as central nervous system tumors, peripheral nerve tumors, epilepsy, Parkinson s disease, movement disorders, Chiari syndrome, central nervous system malformations, and pain disorders)
3. For adults: able to provide informed consent or having a legally-authorized representative to provide consent, if incapacitated
4. For minors: a parent or legal guardian who is able to provide consent.
5. Be willing to consent for collection of clinical data or biological samples or their cryopreservation

3.D. Participant Exclusion Criteria for the cohort with processing of biological samples only (for those subjects who are only having skin biopsies and/or saliva samples)

1. Patients who are unable to undergo evaluation and treatment for a neurosurgical disorder
2. At the time of enrollment, subjects without an established diagnosis of a wellcharacterized disease entity with validated treatment algorithms. In such cases, proposed resource investment, in the opinion of the investigators, would not contribute to further advancement of knowledge

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a variety of neurosurgical disorders who require standard neurosurgical treatment; immediate blood relatives of those subjects in whom genetic testing is performed
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2003-06-04 (Actual)

PRIMARY OUTCOMES:
standard clinical evaluation and treatment | ongoing
  standard clinical evaluation and treatment

CONTACTS AND LOCATIONS:
Overall Officials: John D Heiss, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This study is not a clinical trial. This study design is not compatible with clinical data sharing.

REFERENCES:
- [Derived] Curry BP, Alvarez R, Widemann BC, Johnson M, Agarwal PK, Lehky T, Valera V, Chittiboina P. Robotic Nerve Sheath Tumor Resection With Intraoperative Neuromonitoring: Case Series and Systematic Review. Oper Neurosurg. 2022 Feb 1;22(2):44-50. doi: 10.1227/ONS.0000000000000051. PMID 35007270
- [Derived] Boyle J, Patronas NJ, Smirniotopoulos J, Herscovitch P, Dieckman W, Millo C, Maric D, Chatain GP, Hayes CP, Benzo S, Scott G, Edwards N, Ray Chaudhury A, Lodish MB, Sharma S, Nieman LK, Stratakis CA, Lonser RR, Chittiboina P. CRH stimulation improves 18F-FDG-PET detection of pituitary adenomas in Cushing's disease. Endocrine. 2019 Jul;65(1):155-165. doi: 10.1007/s12020-019-01944-7. Epub 2019 May 6. PMID 31062234
- [Derived] Saldarriaga C, Lyssikatos C, Belyavskaya E, Keil M, Chittiboina P, Sinaii N, Stratakis CA, Lodish M. Postoperative Diabetes Insipidus and Hyponatremia in Children after Transsphenoidal Surgery for Adrenocorticotropin Hormone and Growth Hormone Secreting Adenomas. J Pediatr. 2018 Apr;195:169-174.e1. doi: 10.1016/j.jpeds.2017.11.042. Epub 2018 Feb 1. PMID 29395172
- [Derived] Chatain GP, Patronas N, Smirniotopoulos JG, Piazza M, Benzo S, Ray-Chaudhury A, Sharma S, Lodish M, Nieman L, Stratakis CA, Chittiboina P. Potential utility of FLAIR in MRI-negative Cushing's disease. J Neurosurg. 2018 Sep;129(3):620-628. doi: 10.3171/2017.4.JNS17234. Epub 2017 Oct 13. PMID 29027863
- [Derived] Lu J, Chatain GP, Bugarini A, Wang X, Maric D, Walbridge S, Zhuang Z, Chittiboina P. Histone Deacetylase Inhibitor SAHA Is a Promising Treatment of Cushing Disease. J Clin Endocrinol Metab. 2017 Aug 1;102(8):2825-2835. doi: 10.1210/jc.2017-00464. PMID 28505327
- [Derived] Yong RL, Wu T, Mihatov N, Shen MJ, Brown MA, Zaghloul KA, Park GE, Park JK. Residual tumor volume and patient survival following reoperation for recurrent glioblastoma. J Neurosurg. 2014 Oct;121(4):802-9. doi: 10.3171/2014.6.JNS132038. Epub 2014 Jul 25. PMID 25061868
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-N-0164.html